CLINICAL TRIAL: NCT06055322
Title: Reducing Suicide Risk Among Aging Caregivers of Persons With AD/ADRD: Adapting, Implementing, and Evaluating Dialectical Behavior Therapy Skills Training Interventions
Brief Title: Reducing Suicide Risk Among Aging Caregivers of Persons With AD/ADRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TexasTechU4
Record Dates: First submitted 2023-09-12; First posted 2023-09-26 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Suicide; Depression; Caregiver Burden; Physical Health; Inflammation
Keywords: Suicide Ideation; Older Adults; Family Caregivers; Alzheimer's Disease and Alzheimer's Disease Related Dementias; Dialectical Behavior Therapy
MeSH Terms: conditions — Suicide; Depression; Caregiver Burden; Inflammation; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Adapted Dialectical Behavior Therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted Dialectical Behavior Therapy (Experimental): Adapting Dialectical Behavior Therapy to focus on reducing suicide ideation for family caregivers of persons with AD/ADRD
  Interventions: Behavioral: Adapted Dialectical Behavior Therapy

INTERVENTIONS:
Behavioral: Adapted Dialectical Behavior Therapy — DBT includes skills training groups, unlike other suicide-specific treatments, with modules on distress tolerance, emotion regulation, interpersonal effectiveness, and mindfulness (Linehan, 2014)

SUMMARY:
This project aims to adapt, implement, and evaluate a Dialectical Behavior Therapy skills training group intervention for aging adult family caregivers of person with Alzheimer's Disease and Alzheimer's Disease Related Dementias (AD/ADRD) to reduce suicidality. By adapting this modality, the investigators will provide a scalable intervention tailored for this high-risk population, maximizing the public health impact and improving suicide prevention.

DETAILED DESCRIPTION:
Family caregivers of persons with Alzheimer's Disease and Alzheimer's Disease Related Dementias (AD/ADRD) experience caregiving-related distress and have about 650% higher rates of suicide ideation (SI; 32.32%) compared to the general population (4.3%). Dialectical Behavior Therapy (DBT), an evidence-based intervention for suicide, addresses multiple areas of psychosocial functioning. Standard DBT is often too re-source-intensive (6 months to 1 year of weekly individual sessions and 1.5-2.5-hour weekly skills training group sessions) and is not tailored to family caregivers of persons with AD/ADRD with SI, creating a significant barrier to SI treatment. The investigators will develop, implement, and evaluate an adapted DBT skills training groups tailored to the unique experiences and needs of family caregivers of persons with AD/ADRD to reduce suicide-related out-comes most effectively. Our specific aims are: (1) Adapt DBT skills groups for family caregivers (of persons with AD/ADRD) endorsing direct or indirect SI (directly stated SI vs. indirect indicators of SI) to ensure it applies to direct and indirect SI and considers SI underreporting; (2) Evaluate the feasibility, acceptability, and fidelity of the adapted DBT skills groups in this sample; (3) Assess preliminary effectiveness indicators of the adapted DBT skills groups. For Aim 1, a panel of experts and two stakeholders (Garrison Institute on Aging (GIA) staff; family caregivers of a person with AD/ADRD), will inform the adaptation of DBT skills training to family caregiv-ers of persons with AD/ADRD and shorten to 16 weekly, 1-hour skills groups sessions, over 4 months. For Aims 2 and 3, the investigators will implement the adapted DBT skills training groups among family caregivers of persons with AD/ADRD with direct/indirect SI at screening while providing respite, all at GIA. The investigators will collect relevant demo-graphic data from family caregivers and family caregiver-reported data about the person with AD/ADRD. Over 18 time points (baseline, following weekly DBT sessions, follow-up), participants will complete self-report assessments targeting DBT fidelity/acceptably, SI (direct and indirect), and suicide risk correlates. The investigators will also record DBT session to monitor fidelity. The investigators will track participant recruitment, group attendance, retention as feasibility metrics. The investigators will also use innovative methodology by collecting inflammation biomarkers and heart rate variability data as an indirect SI assessment. Lastly, the investigators will conduct focus groups after the intervention for addi-tional qualitative acceptability and feasibility data. The investigators will also survey GIA site staff to evaluate their perceived acceptability and feasibility of the intervention at GIA. Our hypotheses are that 1) our adapted DBT skills group will be feasible, acceptable, and maintain DBT fidelity, and 2) SI (direct and indirect), suicide risk factors, and inflammation will decrease, and heart rate variability will increase post intervention. Our expected outcomes are to have a scalable DBT group intervention for family caregivers of persons with ADRD, indications of feasibility and acceptability, and preliminary effectiveness indicators. This work will provide a life-saving suicide prevention approach for family caregivers of persons with AD/ADRD, provide students with multidisciplinary research experiences, and significantly strengthen our university research environment.

ELIGIBILITY:
Inclusion Criteria:

* being age 50 and over (as most informal caregivers of persons with AD/ADRD are 50 or older; AARP, 2020; Chi et al., 2019)
* being the primary informal caregiver
* living with an AD/ADRD-diagnosed patient
* being willing to be prodded for bloodspots
* demonstrating English-fluency
* endorsing a direct or indirect SI/suicide risk
* Eligible individuals will score above clinical cutoffs for SI/suicide risk on at least 1 of 3 measures: the Suicide Behavior Questionnaire-R (SBQ-R; score > 6; Osman et al., 2002), Interpersonal Needs Question-naire (INQ; thwarted belonging score > 35; and perceived burden > 17; Mitchell et al., 2020) or the Geriatric De-pression Scale (GDS; score > 5 Heisel et al., 2005).

Exclusion Criteria:

• Participants with neurocognitive impairment will be excluded (a Mini-Mental State Exam score ≤ 23; Folstein et al., 1975; Kochhann et al., 2010)

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Suicide Cognitions Scale-Revised (SCS-R) | All 18 timepoints
  The SCS-R is a 16-item self-report measure that assesses a variety of beliefs, attitudes, expectations, and perceptions associated with the emergence of suicidal thoughts. Importantly, the SCS-R does not directly ask about suicidal thoughts or behaviors, making it an indirect suicide ideation assessment. Previous studies have found that the SCS-R demonstrates excellent internal consistency (α = .96-.98; Bryan et al., 2021; Moscardini et al., 2020).
Beck Scale for Suicide Ideation (BSSI) | through study completion, an average of 6 months
  The BSSI is a 21-item self-report measure with 19 items to evaluate the current intensity of patients' specific attitudes, behaviors, and plans for suicide, including desire for suicide (suicide ideation) and desire for death generally (death ideation). Two items also assess suicide attempt history and intent during the most recent suicide attempt (if applicable). The BSSI has demonstrated good psychometric properties and has good predictive validity for suicide death (Beck et al., 1997; Brown et al., 2000), including among aging adults (Witte et al., 2006).

SECONDARY OUTCOMES:
Interpersonal Needs Questionnaire (INQ) | through study completion, an average of 6 months
  The INQ is a 15-item self-report assessment of thwarted belonging (9 items; scores range from 9 to 63) and perceived burden (6 items; scores range from 6 to 42). The INQ has demonstrated strong psychometric properties, including construct validity among psychiatric outpatients and aging adults (Hill et al., 2015; Van Orden et al., 2012) and strong internal consistency thwarted belonging (.91) and perceived burden (.94; Mitchell et al., 2020).
Geriatric Depression Scale (GDS) | through study completion, an average of 6 months
  The GDS-15 is a 15-item self-report measure of depression, includes a 5-item subscale to assess for suicide ideation, and has been used as a screener for suicide ideation (Cheng et al., 2010). The GDS has been found to have good internal consistency when used with informal caregivers of patients with AD/ADRD (α = .73).
Difficulty in Emotion Regulation Scale (DERS) | through study completion, an average of 6 months
  The DERS is an 18-item, six-subscale self-report measure of emotion regulation. The subscales assess respondents' acceptance of emotions, ability to engage in goal-directed behavior when distressed, impulse control, awareness of emotions, access to strategies for regulation, and clarity of emotions. The DERS-18 subscales have demonstrated good internal consistency (α = .77-.90).
The Distress Tolerance Scale (DTS) | through study completion, an average of 6 months
  The DTS is a 15-item self-report measure of the degree to which individuals experience negative emotions as intolerable. The DTS has demonstrated good internal consistency (α = .91; Anestis et al., 2007).
Interpersonal Sensitivity Scale (INT) | through study completion, an average of 6 months
  The INT is a 10-item self-report measure that assesses participants' abilities to manage relationships via processes associated with interpersonal effectiveness. The INT has demonstrated good internal consistency (α = .91; Lenz et al., 2016).
The Mindful Attention Awareness Scale (MAAS) | through study completion, an average of 6 months
  The MAAS is a 15-item single-dimension self-report measure of trait mindfulness, measuring the frequency of open and receptive attention to and awareness of ongoing events and experience. MAAS has demonstrated good internal consistency (α = .89-.93; Black et al., 2012), including among aging adults (e.g., Mally & Fiocco, 2016).
DBT Acceptability Measure | through study completion, an average of 6 months
  This is an 8-item self-report measure assessing participants' perceived acceptability of DBT (e.g., I would participate in this intervention again). Questions are analyzed separately to indicate acceptability of the adapted DBT manual.
Zarit Burden Interview (ZBI) | through study completion, an average of 6 months
  The ZBI is a 22-item self-report measure of caregiver burden. It has been validated with informal caregivers of patients with AD/ADRD and has been shown to have good internal consistency (0.83-0.92; Hebert et al., 2000; Bedard et al., 2001) and validity (Hebert et al., 2000).
Short Form Health Survey (SF-12) | through study completion, an average of 6 months
  The SF-12 is a 12-item self-report measure of health and has been validated with aging adults (Jakobsson, 2006). The SF-12 is a commonly used instrument to measure health-related quality of life at various ages. The SF-12 has been shown to be psychometrically valid and reliable (Ware et al., 1996; Ware et al., 1997).
Heart Rate Variability (HRV) | through study completion, an average of 6 months
  HRV will be evaluated using Empatica E4 bands, providing autonomic nervous system arousal data, including heart rate. HRV has been used with aging adults and with informal caregivers in past studies (e.g., Brown et al., 2018; James et al., 2021).
Inflammation Markers | through study completion, an average of 6 months
  CRP and IL-6, Blood for analysis will be collected on filter paper (dried blood spots) Dried blood spots are a non-invasive and low-cost method of collecting blood that involves a finger prick with a lancet and blotting the blood onto filter paper (Miller)

CONTACTS AND LOCATIONS:
Locations (1):
- Garrison Institute on Aging, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will not be providing any individual participant data. It will all be aggregate